CLINICAL TRIAL: NCT02307747
Title: Disruption of Circadian Rhythm and Healthcare-related Infection in Patients With Severe Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014-36; RCAPHM14_0336 (Registry Identifier: APHM)
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Infection
Keywords: infection in ICU
MeSH Terms: conditions — Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- trauma patients (Experimental): Blood samples will be collected every 4 hours during 24 h, between day 2 and day 4 after inclusion
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — Blood samples will be collected every 4 hours during 24 h

SUMMARY:
Circadian rhythms, which play crucial roles in physiology, are emerging as important regulators of specific immune functions. Hospitalization in intensive care unit leads to a deep impairment of circadian rhythm. Infection is a frequent event during ICU hospitalization.

The investigators hypothesis is that in trauma patients the lack of circadian rhythm variations is associated with the occurrence of infection. The primary aim of the study is to assess the circadian variations of plasma Bmal1 in the occurrence of healthcare related infection during the 30 days after inclusion. The secondary aims are to assess the plasma expression of circadian genes (Clock, Cry1, Per3, and Rev-erba), the production of cytokines in plasma, and the concentration of cortisol, according to the occurrence of an infection.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients with an injury severity score > 15, requiring mechanical ventilation for at least 24 h during the first 48 h and an arterial catheter.

Exclusion Criteria:

* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
area under the curve representing the maximal expression of Bmal1 gene during the first 24 h following inclusion | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Coiffard B, Diallo AB, Culver A, Antonini F, Hammad E, Leone M, Mege JL. Exacerbation of circadian rhythms of core body temperature and sepsis in trauma patients. J Crit Care. 2020 Dec;60:23-26. doi: 10.1016/j.jcrc.2020.07.010. Epub 2020 Jul 16. PMID 32731102